CLINICAL TRIAL: NCT02176655
Title: Multi-Center, Double-Blind, Placebo Controlled Pilot Study of VVD-101 for the Treatment of Delayed Alcohol-Induced Headaches
Brief Title: Pilot Study of VVD-101 for the Treatment of Delayed Alcohol-Induced Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: Vivid Pharma Inc. (Industry)
Responsible Party: Principal Investigator, Roger K Cady, MD, CEO, Cady, Roger, M.D.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-001VI
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Delayed Alcohol Induced Headache
Keywords: Delayed Alcohol Induced Headache
MeSH Terms: interventions — Sumatriptan; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VVD-101 (Active Comparator): One sumatriptan succinate 12.5 mg combined with acetylsalicylic acid 325 mg (VVD-101) capsule taken after the onset of a delayed alcohol induced headache.
  Interventions: Drug: VVD-101
- Placebo (Placebo Comparator): One placebo capsule to match taken after the onset of a delayed alcohol induced headache.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVD-101 — All subjects will treat 6 headaches with either VVD-101 or placebo in a randomized order.
  Other Names: sumatriptan succinate 12.5 mg & acetylsalicylic acid 325 mg
  Arms: VVD-101
Drug: Placebo — All subjects will treat 6 headaches with either VVD-101 or placebo in a randomized order.
  Arms: Placebo

SUMMARY:
This study proposes to compare the efficacy of sumatriptan and aspirin to placebo as an acute abortive treatment for delayed alcohol induced headache in adult subjects.

DETAILED DESCRIPTION:
The exploratory study will be conducted at 2 investigational sites. Approximately 26 subjects, 21 years of age and older, with a history of delayed alcohol induced headache, as defined by International Classification of Headache Disorders (ICHD-3 beta) will be enrolled. The study will consist of two visits. Subject participation will last approximately 6 months.

At the screening visit (Visit 1), and before any study procedures, an informed consent will be obtained from the subject. A physical, neurological exam, medication history, and pregnancy test (if appropriate) will be performed. Vital signs will be recorded for all subjects. Subjects will also complete the Simple Screening Instrument for Alcohol and Other Drugs (SSI-AOD).

Subjects scoring greater than 4 (not including items 1 and 15) on the SSI-AOD, at Visit 1, will not be eligible for this study and will be referred to their primary care provider for follow up.

Subjects meeting eligibility criteria will be randomized into 1 of 6 different groups. Each group will receive 3 doses of active drug and 3 doses of placebo in a different order to treat up to 6 delayed alcohol-induced headaches. Study product instructions will be reviewed. A copy of the instructions will be given to the subject. Subjects will be instructed they may take their investigator approved routine rescue medications for headaches 2 hours after taking the study medication if needed. Rescue medication usage and dosage will be recorded on the headache diary. Subjects may take acute headache medications as prescribed; however, this should be recorded on the headache diary. Therapy considered necessary for the subject's welfare may be given at the discretion of the investigator. Routine medications should be maintained on a stable dose and regimen for the duration of the study period.

Subjects will be instructed regarding completion of the online Headache Diary to document treatment response of up to 6 delayed alcohol-induced headaches. Subjects will be provided instructions for completing the Headache Diary. The Headache Diary will be completed during each headache and will document the number of drinks consumed in the last sitting, time of last drink consumed, pain severity, headache symptoms, and hangover symptoms before treatment, time of treatment with study products, pain severity at 30 minutes, 1, 2, and 24 hours following treatment, time of headache resolution, and time of meaningful headache relief. The Headache Diary will also include questions to evaluate subject satisfaction with study product. Subjects must be headache-free for 24 hours before recording the onset of and treating another headache. Subjects will be phoned monthly during the study to assess compliance, continued understanding, and to collect any adverse events.

Visit 2 will occur within 1 week following treatment of a 6th attack or between 180-187 days following Visit 1, whichever occurs first. The medical and medication history will be updated and adverse events will be collected. A urine pregnancy test will be performed if appropriate and vital signs to include weight and height will be performed. Subjects will complete the SSI-AOD. Subjects scoring greater than 4 (not including items 1 and 15) on the SSI-AOD will be referred to their primary care provider for follow up. The Diary will be reviewed and any unused study product and used packaging will be collected. Drug accountability will be performed.

ELIGIBILITY:
Inclusion Criteria:

* male or female 21 years or older.
* able to read, understand, and sign the informed consent.
* currently consume alcohol averaging at least four times per month.
* a negative urine pregnancy test at Visit 1, if female, and of childbearing potential. Note: If of childbearing potential, subject must agree to maintain true abstinence or use (or have their partner use) one of the listed methods of birth control for the duration of the study: hormonal contraceptive, intrauterine device (IUD), condoms, diaphragm, and/or vasectomy. The use of barrier contraceptive (condom or diaphragm) should always be supplemented with the use of a spermicide. Note: To be considered not of childbearing potential, subject must be 6 weeks post-surgical bilateral oophorectomy, hysterectomy, or bilateral tubal ligation, or postmenopausal for at least one year.
* at least a one year history of delayed alcohol-induced headache after light to moderate alcohol consumption.
* able to differentiate delayed alcohol-induced headache from any other headache they may experience (e.g., tension-type headache).
* able to stay awake for at least 2 hours after treatment following first dose of study product.
* willing to complete the online headache diary and questionnaires.
* concomitant medication dosages approved by the investigator.
* internet access and an email address for completion of online diary and questionnaires.

Exclusion Criteria:

* > 6 migraine attacks per month during the 3 months previous to screening.
* history of receiving partial or complete relief of hangover headaches from 650 mg of aspirin.
* history of basilar, ophthalmoplegic, or hemiplegic migraine, cluster headache, or secondary headaches (such as due to trauma, infection, alterations of homeostasis, eye, nose, throat (ENT) disorders, or psychiatric disorders, cranial or cervical disorders or neuralgias) within the previous year.
* significant alcohol or drug use problems (score > 4 on the Simple Screening Instrument for Alcohol and Other Drugs (SSI-AOD)) or history of treatment or counseling for alcohol or drug abuse and or dependence.
* used acute headache medication including non-prescription medications, 15 or more days per month during the last 3 months.
* pregnant, actively trying to become pregnant, or breastfeeding.
* female of childbearing potential not using adequate contraceptive measures.
* has a history of serotonin syndrome or in the opinion of the investigator is at an increased risk for developing serotonin syndrome with the use of triptans.
* in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or the presence of risk factors including but not limited to hypertension, hypercholesterolemia, smoker, obesity, diabetes, or family history of coronary artery disease).
* if female, has migraine with aura, is a smoker, and currently taking estrogen containing birth control pill, and in the investigator's opinion, is at high risk for cerebrovascular disease.
* uncontrolled hypertension (≥140/90 mmHg in either systolic or diastolic in 2 out of 3 blood pressure measurements at screening).
* history of any clinically significant medical or psychiatric condition, or evidence of substance abuse including binge drinking within the last year that, in the opinion of the investigator, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this study.
* has hypersensitivity, intolerance, or contraindication to the use of any triptan or aspirin (including all sumatriptan and aspirin preparations).
* has history of nasal polyps and/or asthma and in the investigator's opinion is at risk for hypersensitivity to aspirin.
* participated in an investigational drug trial within the past 30 days.
* planning or requiring surgery during the study.
* history of poor compliance with medical treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - South Drive Medical Clinic, Mountain View, California
  - Clinvest, Springfield, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Sumatriptan succinate 12.5 mg/acetylsalicylic acid 325 mg: All subjects will treat 6 headaches with either VVD-101 or placebo in a randomized order.
  One sumatriptan succinate 12.5 mg combined with acetylsalicylic acid 325 mg (VVD-101) capsule or one placebo capsule to be taken after the onset of a delayed alcohol induced headache.
Period: Overall Study
Arm/Group | All Study Participants
Started | 31
Completed | 25
Not Completed | 6
Not completed — Subjects did not treat | 6

BASELINE CHARACTERISTICS:
Population: All subjects randomized to treatment are included in the baseline analysis population, whether or not they treated a headache.
Groups:
- Cross-Over Group: Sumatriptan succinate 12.5 mg/acetylsalicylic acid 325 mg: All subjects will treat 6 headaches with either VVD-101 or placebo in a randomized order.
  One sumatriptan succinate 12.5 mg combined with acetylsalicylic acid 325 mg (VVD-101) capsule or one placebo capsule to be taken after the onset of a delayed alcohol induced headache.
Arm/Group | Cross-Over Group
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.19 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Headache Severity 2 Hours Post Treatment
Description: Headache severity 2 hours post treatment in sumatriptan succinate 12.5 mg and acetylsalicylic acid 325 mg (VVD-101) vs. placebo. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Prior to Treatment through 2 Hours Post Treatment
Population: Given the design of the study, all subjects treated headaches 1-6 in a randomized fashion with either VVD-101 or placebo, therefore the same 25 subjects are in the VVD-101 and Placebo analysis population. A total of 25 subjects were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VVD-101: One sumatriptan succinate 12.5 mg combined with acetylsalicylic acid 325 mg (VVD-101) capsule taken after the onset of a delayed alcohol induced headache.
  Sumatriptan succinate 12.5 mg/acetylsalicylic acid 325 mg: All subjects will treat 6 headaches with either VVD-101 or placebo in a randomized order.
- Placebo: One placebo capsule to match taken after the onset of a delayed alcohol induced headache.
  Placebo
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre-Treatment | 2.18 (0.63) | 2.09 (0.54)
  2 Hours Post-Treatment | 0.85 (0.88) | 1.17 (0.88)

2. Secondary Outcome: Headache Severity at Treatment, 30 Minutes and 1 Hour Post Treatment
Description: Change in headache severity from before treatment, at 30 minutes, and 1 hour post treatment in attacks treated with VVD-101 vs. placebo. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Prior to Treatment through 1 Hours Post Treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  Pre-Treatment | 2.18 (0.63) | 2.09 (0.54)
  30 Mintues Post-Treatment | 1.78 (0.76) | 1.85 (0.74)
  1 Hour Post-Treatment | 1.20 (0.90) | 1.55 (0.82)

3. Secondary Outcome: Number of Headaches Relieved
Description: Headache relief from before treatment, at 30 minutes, 1 hour, and 2 hours post treatment in attacks treated with VVD-101 vs. placebo. Headache relief is defined as a headache going from moderate or severe to mild or no headache or mild headache going to no headache. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Prior to Treatment to 2 Hours Post Treatment
Population: Given the design of the study, all subjects treated headaches 1-6 in a randomized fashion with either VVD-101 or placebo, therefore the same 25 subjects are in the VVD-101 and Placebo analysis population. A total of 25 subjects, with 87 headaches were analyzed for this endpoint.
Measure: Number; unit: Headaches
Units Other Than Participants: Headaches
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
Number analyzed (Headaches) | 40 | 47
Headaches
  30 Minutes Post-Treatment | 10 | 12
  1 Hour Post-Treatment | 23 | 17
  2 Hours Post-Treatment | 30 | 27

4. Secondary Outcome: Number of Headaches Relieved to Complete Pain Freedom at Two Hours Post Treatment
Description: Number of headaches relieved (no head pain) at 2 hours post treatment for VVD-101 vs. placebo. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Prior to Treatment to 2 Hours Post Treatment
Population: as for outcome 3
Measure: Number; unit: Headaches
Units Other Than Participants: Headaches
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
Number analyzed (Headaches) | 40 | 47
Headaches | 15 | 13

5. Secondary Outcome: Number of Headaches With Sustained Pain Freedom at Twenty Four Hours Post Treatment
Description: Number of headaches with sustained headache pain freedom at 24 hours post treatment for VVD-101 vs. placebo. Sustained headache pain freedom is defined as no pain 2 hours post treatment and headache freedom continuing for 24 hours post treatment without rescue. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Time of Treatment to 24 Hours Post Treatment
Population: Given the design of the study, all subjects treated headaches 1-6 in a randomized fashion with either VVD-101 or placebo, therefore the same 25 subjects are in the VVD-101 and Placebo analysis population. A total of 25 subjects, with 28 headaches were analyzed for this endpoint.
Measure: Number; unit: Headaches
Units Other Than Participants: Headaches
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
Number analyzed (Headaches) | 16 | 12
Headaches | 15 | 12

6. Secondary Outcome: Number of Participants With Consistent Response to VVD-101
Description: To assess the consistency of response to VVD-101 over the three active treatments of VVD-101. Consistency is defined as meeting the requirements of headache relief 2 hours post treatment for 2 out of 3 active treated headaches. Headache relief is defined as a headache going from moderate or severe to mild or no headache or mild headache going to no headache. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Response to Treatment of Three Headaches (estimated 6 months)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VVD-101
Number analyzed (Participants) | 25
participants | 9

7. Secondary Outcome: Satisfaction
Description: To assess subject satisfaction with treatment results comparing VVD-101 vs. placebo. Satisfaction was measured on a 7 point Likert scale whereas 0 = extremely dissatisfied and 6 = extremely satisfied.
Time Frame: 24 Hours Post Treatment for 3 Headaches (estimated 6 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale | 3.75 (2.01) | 2.62 (2.12)

8. Secondary Outcome: Acute Hangover Scale Compared to Pain Severity 2 Hours Post Treatment
Description: Comparison of Acute Hangover Scale (AHS) score before treatment with headache pain severity 2 hours post treatment for headaches treated with VVD-101. The AHS scale is rated on a score of 0-63. A score of 0 indicates no symptoms and a total score of 63 indicates the maximum number of reported symptoms. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Before Treatment of 3 Headaches to 2 Hours Post Treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVD-101
Number analyzed (Participants) | 25
units on a scale
  Acute Hangover Scale Before Treatment | 22.98 (11.82)
  Headache Pain Severity 2 Hours Post Treatment | .85 (.88)

9. Other Pre Specified Outcome: Number of Drinks Consumed Compared to Pain Severity 2 Hours Post Treatment
Description: Comparison of the number of drinks consumed at one sitting with pain severity 2 hours post treatment for headaches treated with VVD-101. Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Time of Last Sitting to 2 Hours Post Treatment (estimated 14 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Drinks Consumed
Arm/Group | VVD-101
Number analyzed (Participants) | 25
Number of Drinks Consumed | 4.71 (2.61)

10. Other Pre Specified Outcome: Comparing Acute Hangover Scale Individual Symptoms With Headache Severity 2 Hours Post Treatment
Description: Comparison of headache severity 2 hours post treatment of headache treated with VVD-101 with each associated hangover symptom items on the AHS taken before treatment. Individual Hangover Symptoms Scores range from 0 [None] to 7 [Incapacitating]. The AHS scale is rated on a score of 0-63. A score of 0 indicates no symptoms and a total score of 63 indicates the maximum number of reported symptoms.Headache severity was measured on a 4 point Likert scale with 0 = no pain, 1 = mild pain, 2 = moderate, 3 = severe pain.
Time Frame: Immediately Before Treatment to 2 Hours Post Treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | VVD-101
Number analyzed (Participants) | 25
units on a scale
  Hangover | 3.53 (1.72)
  Thirsty | 3.5 (1.9)
  Tired | 3.78 (1.54)
  Headache | 4.23 (1.47)
  Dizziness or Faintness | 1.65 (1.77)
  Nausea | 1.75 (1.83)
  Stomach Ache | 1.58 (2.01)
  Heart Racing | 1.10 (1.30)
  Loss of Appetite | 1.88 (1.86)
  Headache Pain Severity 2 Hours Post Treatment | .85 (.88)

11. Other Pre Specified Outcome: Meaningful Headache Relief
Description: Time to meaningful headache relief for VVD-101 vs. placebo. Meaningful headache relief is defined as experiencing substantial relief as reported by the subject.
Time Frame: Time of Onset to Meaningful Headache Relief (up to 24 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | VVD-101 | Placebo
Number analyzed (Participants) | 25 | 25
minutes | 226.33 (268.98) | 351.14 (403.01)

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=31)
Cold (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No